CLINICAL TRIAL: NCT02859285
Title: Sexual Function in Postmenopausal Women: A Double Blinded, Randomized Pilot Study Evaluating the Effects of Topical Clitoral Estradiol Cream
Brief Title: A Study Evaluating the Effects of Topical Clitoral Estradiol Cream in Post Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProHealth Care, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB # 15-18
Record Dates: First submitted 2016-04-20; First posted 2016-08-09 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Arousal; Orgasm; Clitoral; Estradiol; Post Menopausal
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Orgasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol vulvar cream (Active Comparator): The estradiol cream 0.5 grams will be placed on the clitoris/vestibule every night for 2 weeks, then 3 times a week thereafter on Monday, Wednesday, and Friday, for a total of 12 weeks.
  In addition estradiol 10mcg tablet will be placed in the vaginal every night for 2 weeks, then 2x a week on Tuesday and Thursday, for a total of 12 weeks.
  Interventions: Other: Estradiol vulvar cream
- Placebo cream (Placebo Comparator): The placebo cream 0.5 grams will be placed on the clitoris/vestibule every night for 2 weeks, then 3 times a week thereafter on Monday, Wednesday, and Friday, for a total of 12 weeks.
  In addition estradiol 10mcg tablet will be placed in the vaginal every night for 2 weeks, then 2x a week on Tuesday and Thursday, for a total of 12 weeks.
  Interventions: Other: Placebo vulvar cream

INTERVENTIONS:
Other: Placebo vulvar cream
  Arms: Placebo cream
Other: Estradiol vulvar cream
  Arms: Estradiol vulvar cream

SUMMARY:
The purpose of this research study is to learn about sexual function in postmenopausal women and to determine whether the use of topical clitoral application of estradiol improves women's libido, arousal, and orgasmic ability.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active postmenopausal women of any age with complaint of vulvar and/or vaginal atrophy who also complain of bothersome decreased libido, and/or arousal, and/or orgasmic dysfunction

Exclusion Criteria:

* Not sexually active with a partner or an arousal device
* Uncontrolled diabetes as defined by having a consistent blood sugar level of over 100 mg/dL
* Uncontrolled hypertension as defined by an average systolic blood pressure ≥140 mmHg or an average diastolic blood pressure ≥90 mmHg, among those with hypertension
* Allergic to estradiol
* Contraindications to estradiol such as undiagnosed abnormal genital bleeding; known/suspected or history of breast cancer; known/suspected estrogen-dependent neoplasm; active deep vein thrombosis, pulmonary embolism; active or recent stroke or myocardial infarction; liver dysfunction or disease
* Spanish speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2019-03-18 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
19 point validated Female Function Index. | Baseline then change over time at week 4,8,12

SECONDARY OUTCOMES:
36 point RAND health survey. | Baseline then change over time at week 4,8,12.

OTHER OUTCOMES:
10 point Likert scale | Baseline then change over time at week 4,8,12.
  Visual Analog Scale to measure improvement in libido, arousal and orgasm.

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Aschkenazi, MD, Study Director — ProHealth Care, Inc
Locations (1):
- Waukesa Memorial Hospital, Waukesha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided